CLINICAL TRIAL: NCT06132165
Title: Efficacy of Skin Cooling in Reducing Pain Associated With Non-invasive Treatments of Neurofibromatosis Type 1 Cutaneous Neurofibromas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director, Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023P002152
Record Dates: First submitted 2023-11-01; First posted 2023-11-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Deoxycholic Acid; Polidocanol; Lasers, Solid-State

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Kybella Injection (Active Comparator)
  Interventions: Drug: Deoxycholic Acid
- Asclera Injection (Active Comparator)
  Interventions: Drug: Polidocanol
- 1064nm laser (Active Comparator)
  Interventions: Device: 1064nm Nd:YAG laser
- 755nm laser (Active Comparator)
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Drug: Deoxycholic Acid — Injection into the cutaneous Neurofibromas lesion.
  Other Names: Kybella
  Arms: Kybella Injection
Drug: Polidocanol — Injection into the cutaneous Neurofibromas lesion.
  Other Names: Asclera
  Arms: Asclera Injection
Device: 1064nm Nd:YAG laser — Pulse laser at a wavelength of 1064nm to the cutaneous Neurofibromas lesion.
  Arms: 1064nm laser
Device: 755nm Alexandrite Laser — Pulse laser at a wavelength of 755nm to the cutaneous Neurofibromas lesion
  Arms: 755nm laser

SUMMARY:
This study will evaluate the effectiveness of skin cooling in increasing tolerability of four treatments in Neurofibromatosis Type 1 Cutaneous Neurofibromas. These treatments are: a 980nm laser, a 755nm laser, radio-frequency injection, and a Kybella injection. Each patient will have a treatment and a control site..

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. Have a diagnosis of NF1 based on germline genetic testing or by meeting ≥ 2 the following criteria:

   1. Family history of NF1
   2. Six or more light brown ("cafe-au-lait") spots on the skin
   3. Presence of two or more neurofibromas of any type, or one or more plexiform neurofibromas
   4. Freckling under the arms or in the groin area
   5. Two or more pigmented, benign bumps on the eye's iris (Lisch nodules)
   6. A distinctive bony lesion: dysplasia (abnormal growth) of the sphenoid bone behind the eye, or dysplasia of long bones, often in the lower leg
   7. Tumor on the optic nerve that may interfere with vision
3. Patients must be seeking treatment for cNF
4. Patients must have ≥ 6 paired cNF (3 to be treated and 3 untreated) that are visible and measure between 2-8mm in size. These must be in areas amenable to treatment and surveillance with digital photography.
5. cNF must be located on the trunk, arms or legs of the patient
6. Able and willing to comply with all visit, treatment and evaluation schedules and requirements
7. Able to understand and provide written informed consent

Exclusion Criteria:

1. Individuals who cannot give informed consent or adhere to study schedule.
2. Actively tanning during the course of the study.
3. Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
4. Known allergy to injectable anesthetics, deoxycholic acid or polidocanol.
5. Women who are pregnant.
6. Those with acute thromboembolic diseases.
7. Those with bleeding abnormalities or those who are currently being treated with antiplatelet or anticoagulant therapy.
8. Those with dysphagia.
9. Any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months after treatment
  Device based treatment will be considered tolerable if <40% of participants treated have a >grade 2 adverse event (AE). A grade 2 AE is defined as an event that requires treatment.

SECONDARY OUTCOMES:
Patient Report Outcomes | For the 12 months after treatment
  Using questionnaires, we will determine the patients' reported outcomes.
Clinician Reported Outcomes | For the 12 months after treatment
  Using questionnaires we will determine the clinicians' reported outcomes.

OTHER OUTCOMES:
Rate of healing | Baseline, 3 months, 6 months, and 12 months, post-treatment
  Measured by photography completed by member at medical team
cNF Appearance | Baseline, 3 months, 6 months, and 12 months, post-treatment
  Measured via clinically completed 2D and 3D photography

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Boston, Massachusetts, United States